CLINICAL TRIAL: NCT01558635
Title: Evaluation of the Cardioblate CryoFlex Surgical Ablation System in Subjects With Longstanding Persistent Atrial Fibrillation Requiring Mitral Valve Surgery
Brief Title: Evaluation of the Cardioblate CryoFlex Surgical Ablation System in Longstanding Persistent Atrial Fibrillation
Acronym: CRYO-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prematurely closed due to ongoing challenging enrollment requirements.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT-CRYO-001
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Longstanding Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Surgical Ablation; Maze Procedure; AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardioblate CryoFlex Surgical Ablation (Experimental): Subjects with longstanding persistent AF undergoing Maze III procedure using the Cardioblate CryoFlex Surgical Ablation System concomittant to Mitral valve surgery. During surgery, a Medtronic Reveal XT Insertable Cardiac Monitor was implanted to monitor future episodes of AF.
  Interventions: Device: Cardioblate CryoFlex Surgical Ablation; Procedure: Mitral Valve surgery; Device: Medtronic Reveal XT Insertable Cardiac Monitor; Procedure: MAZE III

INTERVENTIONS:
Device: Cardioblate CryoFlex Surgical Ablation — Longstanding persistent AF was treated with the Cox Cryo Maze III procedure During mitral valve surgery a surgical ablation was performed, using the Cardioblate CryoFlex Surgical Ablation System. In addition, the Medtronic Reveal XT Insertable Cardiac Monitor, was implanted.
Procedure: Mitral Valve surgery — Classic mitral valve surgery was performed
Device: Medtronic Reveal XT Insertable Cardiac Monitor — During the procedure, a Medtronic Reveal XT Insertable Cardiac Monitor was implanted to monitor episodes of AF during follow-up period
Procedure: MAZE III — Longstanding persistent AF was treated with the Cox Cryo Maze III procedure

SUMMARY:
Studies have shown that taking drugs to stay out of AF has limited success. This research is designed to study heart rhythm after surgical therapy, namely by measuring if there are benefits to having surgery to treat Atrial Fibrillation (AF) with the Cardioblate CryoFlex Surgical Ablation System. The system is approved and commercially available with CE mark. The purpose of this study is to support clinical evidence that the Cardioblate System is safe and effective to treat AF.

DETAILED DESCRIPTION:
Introduction: Among the cardiac arrhythmias, Atrial Fibrillation (AF) is the most common sustained cardiac arrhythmia in the general population and represents an increasing problem worldwide. Management strategies for AF include combinations of various treatments, including surgery. Cox et al. developed the surgical Maze procedure to restore sinus conduction to the AV node and to restore effective, synchronized bi-atrial contraction. In an effort to address the observed challenges and make this treatment available to more subjects, modifications of the Maze pattern and new lesion patterns have being developed and tested. Devices using new technologies, like cryothermia, were developed in an effort to reduce the time required to make the lesion pattern.The Cardioblate® CryoFlex™ Surgical Ablation System has been successfully used for the surgical ablation of cardiac arrhythmias including atrial fibrillation. The system utilizes cryothermia to create the linear lesions of the surgical Maze-III procedure.

Purpose: To provide clinical evidence showing that the Cox Cryo Maze III procedure is effective and safe in subjects with longstanding persistent AF undergoing mitral valve repair or replacement.

Study objective: The study objectives were to characterize the safety and efficacy of the Medtronic Cardioblate CryoFlex Surgical Ablation System when used to treat subjects with longstanding persistent AF requiring concomitant mitral valve repair or replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented history of longstanding persistent AF as defined by the HRS/EHRA/ECAS Guidelines
* Patients should have a concomitant indication (other than AF) for open-heart surgery for mitral valve repair or replacement (bioprosthesis)
* Patients should be older than or equal to 18 years of age

Exclusion Criteria:

* Atrioventricular reentrant tachycardia (AVRT)
* NYHA Class = IV
* Left ejection fraction of ≤ 30%
* Need for emergent cardiac surgery (i.e. cardiogenic shock) or redo open heart surgery
* Previous atrial fibrillation ablation, AV-nodal ablation, or surgical Maze procedure
* Contraindication for anticoagulation therapy
* Left atrial diameter > 7.0 cm
* Preoperative need for intra-aortic balloon pump or intravenous inotropes
* Renal failure requiring dialysis or hepatic failure
* Life expectancy of less than one year
* Pregnancy or desire to be pregnant within 12 months of the study treatment
* Current diagnosis of active systemic infection
* Documented MI 6 weeks prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vang, MD, Study Director — Medtronic
Locations (4):
- Herzzentrum Leipzig GmbH, Leipzig, Germany
- Sheba Medical Center, Tel Litwinsky, Israel
- San Raffaele Hospital, Milan, Italy
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardioblate CryoFlex Surgical Ablation: Subjects with longstanding persistent AF undergoing Maze III procedure using the Cardioblate CryoFlex Surgical Ablation System concomittant to mitral valve surgery
  Maze III procedure with Cardioblate CryoFlex Surgical Ablation System: During planned mitral valve surgery, longstanding persistent AF was treated with the Cox Cryo Maze III procedure by using Cardioblate CryoFlex Surgical Ablation System. In addition, the Medtronic Reveal XT Insertable Cardiac Monitor, was implanted.
Period: Overall Study
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Started | 17
Treated | 17
Discharge /1 Month Post-procedure | 15
3 Months Post-procedure | 14
6 Months Post-procedure | 14
Completed (12 months post-procedure) | 11
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Subject received other treatment | 1
Not completed — Reveal XT was explanted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
NYHA Class [Count of Participants; unit: Participants] — NYHA I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea. NYHA II: slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). NYHA III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. NYHA IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA Class I | 3
    NYHA Class II | 11
    NYHA Class III | 3
    NYHA Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage of Treated Subjects Diagnosed With Longstanding Persistent AF Off Class I or III Antiarrhythmic Drugs and Out of AF at 12 Months, and Who Did Not Receive Additional Ablation Therapy for AF Prior to the 12-month Evaluation.
Description: The primary efficacy endpoint was defined as the percentage of subjects diagnosed with longstanding persistent AF off Class I or III antiarrhythmic drugs and out of AF, as determined by Reveal XT recordings (AF burden < 0.5% per 24h) at 12 months and who did not receive additional ablation therapy for AF prior to the 12-month evaluation. An additional ablation therapy could include percutaneous catheter ablation or AV nodal ablation (cauterizing or freezing the AV node). Cardioversions were allowed only during the 12 week blanking period.
Time Frame: 12 months
Population: There were 11 subjects with data at 12 months, including antiarrhythmic drug, ablation, and cardioversion data. However, only six subjects had the AF burden data required for the primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 6
Participants | 5

2. Primary Outcome: Safety: Rate of Device and Procedure Related Acute Major Adverse Events (MAE) Within 30 Days Post-procedure or Prior to Hospital Discharge, Whichever Came Last
Description: The composite MAE was defined as a subject experiencing any of the following adverse events:
  * Stroke
  * Transient ischemic attack (TIA)
  * Pulmonary embolism
  * Peripheral arterial embolism
  * Myocardial infarction (MI)
  * Mediastinitis
  * Esophageal injury
  * Death
  * Cardiac injury related to the use of the Cardioblate CryoFlex System that required additional surgical or catheter intervention
Time Frame: 30 days
Population: All subjects treated with the Cardioblate Cryoflex Surgical Ablation System.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 17
Participants
  Cardiac Death | 0
  Non-Cardiac Death | 0
  Stroke | 0
  Transient Ischemic Attack | 1
  Pulmonary Embolism | 0
  Peripheral Arterial Embolism | 0
  Myocardial Infarction | 0
  Mediastinitis | 0
  Esophageal Injury | 0
  Cardiac Injury related to the use of Ablation | 0

3. Secondary Outcome: Number of Participants With Freedom From AF Regardless of Use of Anti-Arrhythmic Drugs
Time Frame: 12 Months
Population: All subjects who underwent ablation therapy and who had data from the Reveal XT Insertable Cardiac Monitor
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Number of Participants With Freedom From AF Regardless of Use of Anti-Arrhythmic Drugs
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 8
Participants | 4

5. Secondary Outcome: Number of Participants With Freedom From AF Regardless of Use of Anti-Arrhythmic Drugs
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 4
Participants | 3

6. Secondary Outcome: AF Burden in Subjects Diagnosed With Longstanding Persistent AF as Measured by Reveal XT Recordings at 3, 6 and 12 Months
Description: AF burden is defined as percentage of time the patient is in AF during 24 hours.
Time Frame: 3, 6 and 12 Months
Measure: Mean (Standard Deviation); unit: percentage of AF burden
Groups:
- AF Burden in Treated Subjects After 3 Months Follow-Up; AF Burden in Treated Subjects After 6 Months Follow-Up; AF Burden in Treated Subjects After 12 Months Follow-Up: Subjects with longstanding persistent AF undergoing Maze III procedure using the Cardioblate CryoFlex Surgical Ablation System concomittant to mitral valve surgery
  Maze III procedure with Cardioblate CryoFlex Surgical Ablation System: During planned mitral valve surgery, longstanding persistent AF was treated with the Cox Cryo Maze III procedure by using Cardioblate CryoFlex Surgical Ablation System. In addition, the Medtronic Reveal XT Insertable Cardiac Monitor, was implanted.
Arm/Group | AF Burden in Treated Subjects After 3 Months Follow-Up | AF Burden in Treated Subjects After 6 Months Follow-Up | AF Burden in Treated Subjects After 12 Months Follow-Up
Number analyzed (Participants) | 8 | 5 | 6
percentage of AF burden | 3.0 (6.7) | 1.3 (2.8) | 2.4 (5.5)

7. Secondary Outcome: Assessment of Quality of Life as Measured by the SF-12 at Baseline, 6 and 12 Months After the Procedure
Description: The 12-Item Short Form Health Survey (SF-12) is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. Ten summary scores are reported from the SF-12. The scale range for each of the ten subscales is from 0 to 100, with higher scores corresponding to a better outcome. Subjects average unit score (with standard deviation) are reported at baseline, 6 and 12 months. As unit of measure we used units on a scale.
Time Frame: 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Quality of Life of Treated Subjects at Baseline; Quality of Life of Treated Subjects at 6 Months Follow-Up; Quality of Life of Treated Subjects at 12 Months Follow-Up: Subjects with longstanding persistent AF undergoing Maze III procedure using the Cardioblate CryoFlex Surgical Ablation System concomittant to mitral valve surgery
  Maze III procedure with Cardioblate CryoFlex Surgical Ablation System: During planned mitral valve surgery, longstanding persistent AF was treated with the Cox Cryo Maze III procedure by using Cardioblate CryoFlex Surgical Ablation System. In addition, the Medtronic Reveal XT Insertable Cardiac Monitor, was implanted.
Arm/Group | Quality of Life of Treated Subjects at Baseline | Quality of Life of Treated Subjects at 6 Months Follow-Up | Quality of Life of Treated Subjects at 12 Months Follow-Up
Number analyzed (Participants) | 16 | 14 | 10
units on a scale
  Physical Component Summary (PCS) | 38.0 (10.4) | 46.7 (10.0) | 43.4 (9.4)
  Mental Component Summary (MCS) | 47.2 (10.3) | 52.7 (12.0) | 56.1 (9.7)
  Physical Functioning | 36.6 (12.8) | 46.6 (10.6) | 42.7 (11.6)
  Role Physical | 37.3 (13.2) | 45.3 (10.0) | 43.4 (11.9)
  Bodily Pain | 45.3 (13.0) | 50.9 (11.7) | 52.3 (7.2)
  General Health | 36.9 (10.8) | 48.4 (8.7) | 46.7 (9.3)
  Vitality | 49.6 (12.3) | 53.5 (11.0) | 54.8 (6.8)
  Social Functioning | 43.9 (13.0) | 50.8 (9.5) | 49.5 (9.6)
  Role Emotional | 39.0 (14.5) | 47.3 (12.4) | 51.0 (7.7)
  Mental Health | 46.6 (10.1) | 53.2 (11.7) | 54.8 (10.0)

8. Secondary Outcome: Rate of Device and Procedure Related Acute Major Adverse Events (MAE) Within 12 Months Post-procedure or Prior to Hospital Discharge, Whichever Came Last
Description: as for outcome 2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioblate CryoFlex Surgical Ablation
Number analyzed (Participants) | 17
Participants
  Cardiac Death | 0
  Non-Cardiac Death | 0
  Stroke | 0
  Transient Ischemic Attack (TIA) | 1
  Pulmonary Embolism | 0
  Peripheral Arterial Embolism | 0
  Mediastinitis | 0
  Esophageal Injury | 0
  Cardiac Injury related to the use of Ablation | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Groups:
- Cardioblate CryoFlex Surgical Ablation Group With 12 Months of: Subjects with longstanding persistent AF undergoing Maze III procedure using the Cardioblate CryoFlex Surgical Ablation System concomittant to Mitral valve surgery
  Maze III procedure with Cardioblate CryoFlex Surgical Ablation System: During planned mitral valve surgery, longstanding persistent AF was treated with the Cox Cryo Maze III procedure by using Cardioblate CryoFlex Surgical Ablation System. In addition, the Medtronic Reveal XT Insertable Cardiac Monitor, was implanted.
Arm/Group | Cardioblate CryoFlex Surgical Ablation Group With 12 Months of
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioblate CryoFlex Surgical Ablation Group With 12 Months of (N=17)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Ventriculr Block, Second Degree (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemodynamic Instability (Vascular disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2)
Bundle Branch Block, Right (Cardiac disorders) | 1 (1)
Haematoma Infection (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular Block, Complete (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioblate CryoFlex Surgical Ablation Group With 12 Months of (N=17)
Arterial Hypotension (Vascular disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Transient Psychosis (Psychiatric disorders) | 2 (2)
Hyponatriaemia (Metabolism and nutrition disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative Delirium (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Anemia (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was prematurely stopped due to sustained difficulties in the recruitment of eligible subjects. As a result only 17 subjects were enrolled in the study. Reveal XT data were retrievable in only 6 of the enrolled subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less